CLINICAL TRIAL: NCT00578903
Title: Allogeneic Stem Cell Transplantation for Patients With Severe Aplastic Anemia, Using Matched Unrelated Donors and Mismatched Related Donors (SAA MUD)
Brief Title: Allogeneic Stem Cell Transplant for Patients With Severe Aplastic Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kathryn Leung, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10915-SAA MUD; SAA MUD; NCT00598221 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Aplastic Anemia
Keywords: Severe Aplastic Anemia; Severe
MeSH Terms: conditions — Anemia, Aplastic; Lymphoma, Follicular | interventions — Cyclophosphamide; Alemtuzumab; Whole-Body Irradiation; Radiation; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Patients with a diagnosis of severe aplastic anemia who require an allogeneic stem cell transplant but lack an Human Leukocyte Antigen (HLA) identical family member.
  Cytoxan, Campath, TBI-Total Body Irradiation, FK-506, Methotrexate, Stem Cell Infusion
  Interventions: Drug: Cytoxan; Drug: Campath; Radiation: Total Body Irradiation (TBI); Drug: FK-506; Drug: Methotrexate; Procedure: Stem cell infusion

INTERVENTIONS:
Drug: Cytoxan — Cytoxan will be given at 50 mg/kg per dose for 4 successive days.
  Other Names: Cyclophosphamide
Drug: Campath — Campath will be given at a dose of 3 mg for patients whose weight is between 5 and 15 kg; at a dose of 5 mg for patients whose weight is between 16 and 30 kg; and at a dose of 10 mg for patients whose weight is greater than 30 kg. The last dose of Campath should be 24 hours or more before stem cell infusion.
  Other Names: alemtuzumab
Radiation: Total Body Irradiation (TBI) — TBI will be given at a dose of 200 cGy for 6/6 HLA match and at a dose of 400 cGy in two fractions of 200 cGy each for 5/6 HLA matched donor.
  Other Names: Irradiation
Drug: FK-506 — FK-506 will be given at a dose of 0.03 mg/kg/day via continuous infusion over 24 hours from 4pm on day -2 until engraftment or when patient is able to take by mouth (PO), then 0.03 mg/kg PO every 12 hours.
  Other Names: Tacrolimus
Drug: Methotrexate — Methotrexate will be administered on day +1, day +3, day +6 and day +11 at a dose of 5 mg/m2. The day +11 dose may be omitted at the discretion of the bone marrow transplant (BMT) in-patient attending physician.
Procedure: Stem cell infusion — Where possible patients will receive bone marrow. Marrow will be collected as per National Marrow Donor Program (NMDP) guidelines to provide a volume of 15-20 ml/kg of marrow and/or 2-4 X 10^8 nucleated cells/kg. In case marrow cannot be collected, peripheral blood stem cell (PBSC) will be substituted. A minimum of 5-6 X 10^6 CD 34+ cells/kg should be collected, with a target of 10 X 10^6/kg.

SUMMARY:
Patients have been diagnosed with severe Aplastic Anemia that have not responded to treatment with immunosuppressive therapy (drugs that suppress the immune system, for example Steroids). The immune system is the system in the body that helps protect the body and fights bacterial, viral and fungal infections.

Research studies have shown that patients with Aplastic Anemia have improved survival (may live longer) after receiving a HLA (Human Leukocyte Antigen) identical sibling (brother and sister) stem cell transplants. Patients who do not have matched siblings can undergo immunosuppressive therapy, which has also shown to improve outcome. Unfortunately patients who do not respond to immunosuppressive therapy usually die. The best chance of survival for these patients is an HLA matched unrelated or mismatched related stem cell transplant as described below.

Stem cells are created in the bone marrow. They mature into different types of blood cells that people need including red blood cells which carry oxygen around the body, white blood cells which help fight infections, and platelets which help the blood to clot and prevent bleeding. For a matched unrelated stem cell transplant, stem cells are collected from a person (donor) who is not related to the patient but who has the same type of stem cells. For a mismatched related stem cell transplant, stem cells are collected from a donor who is related to the patient and whose stem cells are almost the same as those of the patient but not exactly. The patient then receives high dose chemotherapy. This chemotherapy kills the stem cells in the patient's bone marrow. Stem cells that have been collected from the donor are then given to the patient to replace the stem cells that have been killed.

The major problems associated with these types of stem cell transplants are graft rejection (where the patient's immune system rejects the donor stem cells) and severe graft versus host disease (GVHD), where the donors stem cell reacts against the patient's tissues in the body.

DETAILED DESCRIPTION:
Before patients receive any treatments, they will have the following:

* Complete history and physical exam
* Dental consultation
* Bone marrow aspirate
* Blood tests
* Urinanalysis
* Tests to look at your lungs (Chest X-ray and PFT's and DLCO)
* Tests to look at your heart (EKG, MUGA, or echocardiogram)
* Pregnancy test for females of childbearing age.

Once the decision has been made by the patients to have a mismatched related or matched unrelated stem cell transplant, the patient will receive treatment called a "conditioning regimen" to prepare their body for the transplant. The purpose of this conditioning regimen is to kill the stem cells in the bone marrow, so that the patients immune system is suppressed (lowered or stopped from working), so their body will not reject the donors stem cells (transplant).

The medicines which will be given as part of the conditioning regimen include Cyclophosphamide (Cytoxan) and Campath 1H. Both of these medications are approved by the Food and Drug Administration. Cyclophosphamide will be given for four days in a row. Cyclophosphamide is broken down into different chemicals and removed from the body in the urine. These different chemicals can cause bleeding in the bladder. Mesna is a drug that will be given with Cytoxan to prevent the build up of these chemicals that cause bleeding from the bladder. Campath 1H will also be given for four days. After the medicines, the patient will receive total body irradiation (TBI). Total body irradiation is strong doses of radiation (like x-rays) given to almost the whole body. One dose of TBI will be given to patients receiving a matched stem cell infusion while two doses of TBI will be given to patients receiving a mismatch stem cell infusion. After the conditioning regimen, the patient will then receive the stem cells (transplant). These stem cells will be given as an infusion (drip) into a vein.

Patients will receive the drugs Tacrolimus (FK506) and Methotrexate to help prevent the complication of graft versus host disease. Methotrexate will be given on days 1, 3, 6 and 11 after they receive the stem cells. During this time, the patient will be on the stem cell transplant unit in protective isolation to help protect from developing infections.

The following evaluations will be done as part of the stem cell transplant.

EVALUATION DURING THE FIRST 100 DAYS:

* Physical examination daily until discharged, then weekly.
* Peripheral Blood for chimerism studies (looks at the presence of cells from the donor and from the patient existing together after the transplant)
* Complete blood count (CBC) and platelets daily until discharge, then at least weekly
* Blood chemistry (Electrolytes, BUN, creatinine, glucose, calcium, uric acid, total protein, albumin, ALT, AST, LDH, total bilirubin, LDH, magnesium) checked daily until discharge, then at least weekly
* FK506 blood levels twice a week until discharge, then at least weekly
* Blood tests for CMV (a type of virus) weekly

DAY 100-365:

* Physical examination at least monthly through Day 365
* Peripheral blood for chimerism studies
* Follow-up for patients with chronic GVHD as needed
* Chest X-ray
* CBC and Blood chemistry tests as above checked monthly

YEARLY EVALUATION:

* Biopsies as needed (taking tissue samples for testing)
* Chest x-ray
* CBC and Blood chemistry evaluations as listed above
* Peripheral blood for chimerism studies

IMMUNOLOGIC TESTING:

We will also be looking at the patients immune function. To do this, we will take 30 ml (2 tablespoonfuls) of blood every two weeks for two months, then monthly for 6 months, and then every 3 months for 2 years. When possible, the blood that is taken will be taken through an existing IV line. However, at times drawing the blood will require another stick with a needle. These blood tests will be done for research purposes as part of this study. All other blood tests listed above are done as part of good clinical care for patients receiving a stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Severe Aplastic Anemia (SAA) based on bone marrow aspirate and biopsy results.
2. Failure to respond to immunosuppressive therapy.
3. Lack of an Human Leukocyte Antigen (HLA) identical family member.
4. A 6/6 or 5/6 HLA matched unrelated donor or a 5/6 matched related donor available after high resolution HLA typing.
5. Age from birth to 60 years.

Exclusion Criteria:

1. Severe disease other than aplastic anemia that would limit the probability of survival during the graft procedure. Patients who present with active infection must be treated to maximally resolve this problem before beginning the conditioning regimen.
2. Human immunodeficiency virus (HIV) seropositive patients
3. Patients who have clonal cytogenetic abnormalities or a myelodysplastic syndrome.
4. Patient greater than 60 years of age.
5. Women who are pregnant or nursing.
6. Patients with active hepatitis
7. Patients with severe cardiac dysfunction defined as shortening fraction < 25%.
8. Patients with severe renal dysfunction defined as creatinine clearance < 40 ml/mim/1.73m2.
9. Patient with severe pulmonary dysfunction with forced expiratory volume in the first second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLCO) 40% of predicted or 3 standard deviations (SD) below normal.

Ages: 1 Minute to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2002-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Leung, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Diagnosis SAA, failure to respond to immunosuppressive therapy, lack of HLA identical family member, A 6/6 or 5/6 HLA matched unrelated donor or a 5/6 matched related donor available after high resolution typing, age<60 years
Pre-assignment Details: Pirour to initicating the SCT preparatory regimen, patients require a double lumen Hickman catheter and completion of the pretransplant evaluation.
Groups:
- Patients: Patients with a diagnosis of severe aplastic anemia who require an allogeneic stem cell transplant but lack an Human Leukocyte Antigen (HLA) identical family member.
Period: Overall Study
Arm/Group | Patients
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 22
Age, Customized [Number; unit: participants]
  0-10 years | 9
  11-20 years | 12
  21-30 years | 0
  31-40 years | 0
  41-50 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Alive at 100 Days Post Transplant
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 22
participants | 21

2. Secondary Outcome: Number of Patients With Engraftment Rate at 100 Days Post Transplant
Description: Absolute neutrophil count greater than 0.5 X 10^9/ml for at least 3 days
Time Frame: 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 22
participants | 19

3. Secondary Outcome: Number of Patients With Acute GVHD at 100 Days Post Transplant
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 22
participants | 4

4. Secondary Outcome: Number of Patients With Chronic GVHD at 2 Years Post Transplant
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 22
participants | 1

5. Secondary Outcome: Number of Subjects Alive at 1 Year Post Transplant
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 22
participants | 20

6. Secondary Outcome: Number of Subjects Alive at 2 Years Post Transplant
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 22
participants | 20

ADVERSE EVENTS:
Arm/Group | Patients
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Patients (N=22)
Hypertension (Cardiac disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 1 (2)
Catheter-Related Infection (Infections and infestations) | 2 (3)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 1 (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 6 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Neurology-Other (Nervous system disorders) | 1 (1)
Seizure(s) (Nervous system disorders) | 1/11 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=22)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (8)
Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies, if specifi (Skin and subcutaneous tissue disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 6 (11)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 10 (19)
Stomatitis/Pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (29)
Alkaline Phosphatase (Hepatobiliary disorders) | 3 (3)
Bilirubin (Hepatobiliary disorders) | 3 (6)
GGT (Gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 8 (26)
Hypoalbuminemia (Hepatobiliary disorders) | 10 (28)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 10 (29)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 13 (38)
Bicarbonate (Metabolism and nutrition disorders) | 4 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (10)
Hypernatremia (Metabolism and nutrition disorders) | 2 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (9)
Hypokalemia (Metabolism and nutrition disorders) | 12 (56)
Hypomagnesemia (Metabolism and nutrition disorders) | 13 (47)
Hypomagnesmia (Metabolism and nutrition disorders) | 6 (24)
Hyponatremia (Metabolism and nutrition disorders) | 15 (34)
Abdominal pain or cramping (General disorders) | 3 (3)
Headache (General disorders) | 4 (9)
Pain-Other (General disorders) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine (Renal and urinary disorders) | 2 (8)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal/Genitourinary-Other (Renal and urinary disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes